CLINICAL TRIAL: NCT01845792
Title: Phase II Study of Abiraterone Acetate and Prednisone in Combination With Cabazitaxel, Compared to Cabazitaxel Alone, in Patients With Metastatic Castrate Resistant Prostate Cancer.
Brief Title: Study of Abiraterone Acetate and Prednisone in Combination With Cabazitaxel in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1489.cc; NCI-2013-01356 (Other: National Cancer Institute)
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Metastatic Castrate Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabazitaxel with Abiraterone Acetate (Experimental): Cabazitaxel administered as a single intravenous dose every 3 weeks, in combination with abiraterone acetate and prednisone taken daily.
  Interventions: Drug: Cabazitaxel with Abiraterone Acetate
- Cabazitaxel Alone (Active Comparator): Cabazitaxel administered as a single intravenous dose every 3 weeks
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel with Abiraterone Acetate — Cabazitaxel intravenously every 3 weeks, in combination with abiraterone acetate and prednisone orally daily.
  Other Names: Jevtana; Zytiga
  Arms: Cabazitaxel with Abiraterone Acetate
Drug: Cabazitaxel — Cabazitaxel intravenously every 3 weeks
  Other Names: Jevtana
  Arms: Cabazitaxel Alone

SUMMARY:
Patients are being asked to take place in this research study because they have advanced prostate cancer that has gotten worse after other treatments. If they join this study they will receive a new combination of drugs that are used to treat prostate cancer.

DETAILED DESCRIPTION:
Abiraterone acetate and cabazitaxel have been approved by the United States Food and Drug Administration (FDA) to treat prostate cancer that has spread to other parts of the body such as the lymph nodes or bone. These drugs are approved individually for use when the cancer has become resistant to other treatments, including chemotherapy with docetaxel. The combination of these two drugs has not been evaluated, so the research team will study the safety and effectiveness of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained.
* Adults over 18 years of age.
* Histologically or cytologically proven adenocarcinoma of the prostate.
* Stage IV disease as evidenced by soft tissue, visceral and/or bony metastasis must be Response Evaluation Criteria in Solid Tumors (RECIST) evaluable on CT scan and/or bone scan
* Progressive disease while receiving hormonal therapy or after surgical castration documented by at least one of the following:

  1. Increase in measurable disease per RECIST 1.1,
  2. Appearance of new lesions on bone scan consistent with progressive prostate cancer (>2 new lesions on bone scans if this is the only measure of PD),
  3. rising PSA defined as 2 sequential increases above a previous lowest reference value.

     * Each value must be obtained at least 1 week apart.
* PSA at least 2 ng/mL
* Received prior docetaxel chemotherapy
* Received prior abiraterone acetate, but not within the 3 months prior to study drug dosing.
* Testosterone level <50 ng/mL. Patients receiving Leutinizing Hormone Releasing Hormone (LHRH) agonists or antagonists must be continued to maintain castrate levels of testosterone while on study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate hematologic function:

  1. platelet >100, 000/uL;
  2. neutrophil count of >1500 cell/mm3;
  3. hemoglobin >9.0 g/dL)
* Adequate renal function (Creatinine clearance > 50 mL/min)
* Adequate potassium level (> 3.5 mEq/dL)
* Adequate hepatic function

  1. bilirubin < 1.5 X upper limit of normal (ULN),
  2. alanine aminotransferase (ALT) < 1.5 X ULN,
  3. aspartate aminotransferase (AST) < 1.5 X ULN.
  4. serum albumin of ≥ 3.0 g/dL.
* Controlled blood pressure, defined as blood pressure ≤ 140/90 on average (3 separate readings taken at screening visit in a relaxed clinical environment and averaged)
* Must be able to take oral medication without crushing, dissolving or chewing tablets
* Willing to take abiraterone acetate on empty stomach;

  (1) no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken.
* Patients must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
* Written authorization for use and release of health and research study information has been obtained.
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection during the study and for 1 week after the last dose of abiraterone acetate.

Exclusion Criteria:

* Surgery or radiation therapy within 2 weeks, or
* Cytotoxic anti-cancer therapy within 3 weeks, or
* Non-cytotoxic anti-cancer therapy within 2 weeks, or 5 half-lives (whichever is shorter) of Study Day 1.
* Prior radiotherapy to ≥ 40% of bone marrow.
* Prior treatment with Radium 223.
* Use of an investigational therapeutic agent within 30 days.
* Have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents.
* Prior treatment with cabazitaxel.
* Known chronic infection with human immunodeficiency virus (HIV).
* Known active, or symptomatic, brain metastasis.
* Blood pressure >140/90 on average (3 separate readings taken at screening visit in a relaxed clinical environment and averaged).
* History of autoimmune disorder requiring daily corticosteroid therapy of greater than prednisone 10mg daily, or its equivalent.
* Baseline peripheral edema > grade 3.
* Pre-existing diarrhea uncontrolled with supportive care;
* Prior hemorrhagic diarrhea due to ulcerative colitis, inflammatory bowel disease or other cause;
* Active, uncontrolled peptic ulcer disease even in the setting of proton-pump inhibitor or Histamine2-blocker use.
* Pre-existing peripheral neuropathy grade > 2.
* Documented hypersensitivity (CTCAE grade > 2) to any drug containing polysorbate 80.
* Have known allergies or hypersensitivity to abiraterone acetate or prednisone or their excipients.
* Contraindications to steroid use.
* Need for medications that strongly induce or inhibit cytochrome P450 3A4 (CYP3A4) or cytochrome P450 2D6 (CYP2D6) activity. (see section 7.2.3 for details)
* Serious infection requiring parenteral antibiotics within 14 days of enrollment.
* Poorly controlled diabetes (Hgb A1C >9).
* Active or symptomatic viral hepatitis or Chronic liver disease, including Child-Pugh Class B and C liver disease.
* History of pituitary or adrenal dysfunction.
* Clinically significant heart disease as evidenced by:

  1. myocardial infarction, or
  2. arterial thrombotic events in the past 6 months,
  3. severe or unstable angina, or
  4. New York Heart Association Class III-IV heart disease, or
  5. cardiac ejection fraction measurement of <50% at baseline.
* Consumption of food or beverages containing grapefruit juice within 7 days of study drug dosing
* Use of a first-generation anti-androgen such as:

  1. bicalutamide within 6 weeks of study drug dosing, or
  2. flutamide within 4 weeks of study dosing.
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Lam, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabazitaxel With Abiraterone Acetate | Cabazitaxel Alone
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabazitaxel With Abiraterone Acetate | Cabazitaxel Alone | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7
Prior Docetaxel AND Abiraterone [Count of Participants; unit: Participants] | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free survival at 3 months.
Time Frame: 3 months
Population: Due to early closure of the study and the low number of patients enrolled, no statistics or firm conclusions can be made.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabazitaxel With Abiraterone Acetate | Cabazitaxel Alone
Number analyzed (Participants) | 5 | 2
Participants | 5 | 2

2. Secondary Outcome: PSA Response
Description: Prostate specific antigen (PSA) decline by 50% or more from baseline.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cabazitaxel With Abiraterone Acetate | Cabazitaxel Alone
Number analyzed (Participants) | 5 | 2
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: Patients were on study between 3 to 14 months. Adverse event data were collected throughout study.
Description: Due to early closure and small number of patients enrolled, no statistics or firm conclusions can be made. The 5 patients treated in the combination arm were treated with the standard dosing of both abiraterone acetate and cabazitaxel.
Arm/Group | Cabazitaxel With Abiraterone Acetate | Cabazitaxel Alone
All-Cause Mortality (participants affected / at risk) | 5/5 | 2/2
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel With Abiraterone Acetate (N=5) | Cabazitaxel Alone (N=2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 4 Neutropenia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT01845792/Prot_SAP_000.pdf